CLINICAL TRIAL: NCT02725658
Title: Monitoring and Predicting Breast Cancer Neoadjuvant Chemotherapy Response Using Diffuse Optical Spectroscopic Imaging in a Multi-Center Setting
Brief Title: Monitoring and Predicting Breast Cancer Neoadjuvant Chemotherapy Response Using DOSI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study doesn't meet NIH criteria of clinical trial study
Sponsor: Beckman Laser Institute and Medical Center (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Beckman Laser Institute and Medical Center, Bruce Tromberg, PhD, Director Beckman Laser Institute and Medical Clinic, Professor, Departments of Biomedical Engineering and Surgery, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20152355
Record Dates: First submitted 2016-01-29; First posted 2016-04-01 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Breast Tumor
Keywords: Neoadjuvant Therapy; Diffuse Optical Spectroscopic Imaging; DOSI; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DOSI (Other)
  Interventions: Device: DOSI

INTERVENTIONS:
Device: DOSI — Breast tissue properties scanning
  Other Names: Diffuse Optical Spectroscopy

SUMMARY:
The purpose of this research study is to help us learn if an experimental imaging device called Diffuse Optical Spectroscopic Imaging (DOSI) can monitor tumor shrinkage during chemotherapy treatment and can predict if the tumor will respond to chemotherapy before the end of the treatment. This study will also help us understand the biological reason for how DOSI works.

DETAILED DESCRIPTION:
There is considerable interest in developing imaging protocols to monitor and predict breast cancer response to neoadjuvant chemotherapy (NAC), which is chemotherapy given before surgical removal of the tumor, both prior to and as early as possible during the course of treatment. The efficacy and practicality of conventional imaging approaches in the NAC setting varies and identifies the need for alternate functional imaging strategies. Diffuse optical spectroscopic imaging (DOSI) is an experimental imaging method that allows patients to be followed before and during treatment with a cost-effective, bedside, handheld scanning probe. DOSI is a non-invasive technology developed at the University of California, Irvine Beckman Laser Institute. Studies will be performed at seven clinical sites on approximately 200 suspected breast cancer patients, of which 150 are expected to undergo neoadjuvant chemotherapy (NAC).

As a primary aim, the investigators will evaluate whether DOSI can predict NAC pathologic complete response (pCR), which is defined as no tumor cell left in the resected tissue at surgery) by the mid-point of the therapy regimen. As non-invasive DOSI is obtained rapidly with no risk/discomfort, this experimental imaging modality could be used as an indicator of pathologic response which has been an established indicator of long-term survival. The investigators long-term goal is to provide oncologists with a relatively simple, risk-free bedside tool that can be used to help inform medical decisions on chemotherapy regimen, duration, and timing of surgery, thereby maximizing therapeutic response and minimizing unnecessary toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 21 and 80. Specific to Study part #1
* Diagnosed with a Breast Imaging-Reporting and Data System score of 4 or higher breast abnormality greater than 1cm in size Specific to Study part #2
* Enrolled in study part #1
* Diagnosed with histologically-proven invasive breast cancer
* Prescribed neoadjuvant chemotherapy for breast cancer

Exclusion Criteria:

* Pregnant
* Unable to give written, informed consent.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of oxy-hemoglobin (HbO2), in blood. | through study completion, an average of 3 years
Concentration of deoxy-hemoglobin (HHb) in blood. | through study completion, an average of 3 years
Concentration of total hemoglobin in blood. | through study completion, an average of 3 years
Water content of tissue (%) | through study completion, an average of 3 years
Bulk lipid in tissue (%) | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Tromberg, PhD, Principal Investigator — Beckman Laser Institute
Locations (4):
- United States (4):
  - Pacific Breast Care Clinic, Costa Mesa, California
  - Beckman Laser Institute University of California Irvine, Irvine, California
  - University of California, Irvine Medical Center, Irvine, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No